CLINICAL TRIAL: NCT05464797
Title: Diagnostic Biomarkers to Correlate Molecular Changes and Early Inflammatory Cascade in Deep Carious Lesions With Dental Pulp Exposure.
Brief Title: Diagnostic Biomarkers to Correlate Molecular Changes and Inflammatory Cascade in the Dental Pulp.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02031120
Record Dates: First submitted 2022-07-11; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2020-10

CONDITIONS: Vital Pulp Therapy
Keywords: Partial Pulpotomy; Cytokines; Direct Pulp Capping

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Placebo Comparator)
  Interventions: Diagnostic Test: Cytokines level in pulpal blood.
- Direct Pulp Capping group (Experimental)
  Interventions: Procedure: Pulp therapy; Diagnostic Test: Cytokines level in pulpal blood.
- Partial Pulpotomy group (Experimental)
  Interventions: Procedure: Pulp therapy; Diagnostic Test: Cytokines level in pulpal blood.
- Complete Pulpotomy group (Experimental)
  Interventions: Procedure: Pulp therapy; Diagnostic Test: Cytokines level in pulpal blood.
- Root canal treatment group (Experimental)
  Interventions: Procedure: Pulp therapy; Diagnostic Test: Cytokines level in pulpal blood.

INTERVENTIONS:
Procedure: Pulp therapy — partial or complete removal of inflamed pulp tissue
  Arms: Complete Pulpotomy group; Direct Pulp Capping group; Partial Pulpotomy group; Root canal treatment group
Diagnostic Test: Cytokines level in pulpal blood. — Measuring the concentration of IL-8 and MMP-9 in the dental pulp during inflammation.

SUMMARY:
This study aimed to evaluate the molecular changes that occur within the pulp tissue during inflammation and its correlation with vital pulp therapy with its different treatment modalities (Direct pulp capping, Partial Pulpotomy and Complete Pulpotomy).

DETAILED DESCRIPTION:
The diagnosis of irreversible pulpitis was based only on the clinical signs and symptoms which does not always match that of the histological changes of the pulp tissues. So, it is more appropriate to diagnose the pulp according to the molecular changes taking place throughout the pulp tissues. Different studies have been conducted to study the molecular changes that take place in the inflamed pulp, Including a study that was conducted by Rechenberg et al in 2014 which states different locations to obtain samples for these molecules. The best of which was the dental pulp blood sample. Many studies stated the way to obtain a blood sample from the pulp and how to prepare and test it to evaluate the levels and concentrations of different inflammatory molecules. Many studies were also conducted to study the different changes and accurateness of measurement of different molecules.

The pulp inflammation occurs in a low compliance environment of dentinal walls. So, During acute inflammatory reaction, Vasodilatation occurs along with increased capillary permeability, Which leads to increase in the pulp interstitial fluid pressure which creates more pressure on blood vessels and this prevents beneficial blood flow, which decreases the ability of the pulp to defend itself from bacterial attacks causing tissue necrosis. This necrotic tissue is colonized by bacterial tissues.

In the literature, one of the novel treatment modalities for irrevesible inflammation of the pulp is partial removal of the inflammed pulp tissue according to clinical sign (bleeding control), The pulp tissue is removed partially until reaching complete coronal pulp removal or complete pulpectomy until hemostasis is obtained after 10 minutes of moist cotton pellet application.So, The normal pulp is preserved.

In 2019, Ricucci et al conducted a systematic review for treatment of deep carious lesions with pulp exposure. With treatment modalities ranging from direct pulp capping, partial pulpotomy, complete pulpotomy and pulpectomy. Based only on clinical signs of normal appearance of the pulp tissue under magnification with dental operating microscope and bleeding control within 10 minutes with a moist cotton pellet.

ELIGIBILITY:
Inclusion Criteria:

* Positive response to cold testing.
* The age range from 15-45 years.
* Patients of both sex.
* Has clinical symptoms of pulpitis with normal apical tissues and supported by radiographic evaluation with no periradicular changes.

Exclusion Criteria:

* Patients over 45 years of age.
* Patients with clinical symptoms of periradicular inflammation or periradicular radiographic changes.
* Negative response to cold testing.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Periradicular condition of the teeth | 6 months
  Presence of any radiographic abnormal periapical change
Level of Interleukin 8 in pulpal blood | 6 months
  Severity of inflammation

SECONDARY OUTCOMES:
Level of Matrix metalloproteinase 9 in pulpal blood | 6 months
  Cytokines level in pulpal blood

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahliya, Egypt